CLINICAL TRIAL: NCT00847041
Title: Microarray Analysis of Sinus Samples From Patients With and Without Chronic Rhinosinusitis.
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Department of Otolaryngology - Head and Neck Surgery, University of California, San Francisco
Other Study IDs: A109753
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Rhinosinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the bacteria, fungi, and viruses that are present in the sinuses of patients with chronic rhinosinusitis to patients without sinus disease using a new technology, called a microarray, that will allow more accurate identification of microorganisms than current laboratory methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* History of chronic rhinosinusitis (CRS)
* Impaired CRS-specific quality of life
* Evidence of sinus disease on a CT scan

Exclusion Criteria:

* Control patients with any evidence of CRS by history, survey, or imaging criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty total patients are being recruited: ten adult patients who meet the clinical criteria for chronic rhinosinusitis requiring surgical therapy and ten adult patients undergoing either orbital decompression for Graves' orbitopathy or maxillomandibular advancement for obstructive sleep apnea, with no history of sinus disease.
Sampling Method: Probability Sample